CLINICAL TRIAL: NCT06144502
Title: Promoting Mental Health and Wellbeing Through a School-based Intervention - a Study Using a Mixed-methods, Quasi-experimental Extended Selection Cohorts Design
Brief Title: Promoting Wellbeing: The Five Ways at School Intervention
Acronym: 5Ways@School
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moss Kommune (Other Government)
Collaborators: University of Oslo (Other); Norwegian Institute of Public Health (Other Government); Norwegian Council for Mental Health (Other)
Responsible Party: Principal Investigator, Kristian Green Krogshus, MD, District Medical Officer and PhD candidate, Moss Kommune
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 110419; 345560 (Other Grant/Funding Number: The Research Council of Norway)
Record Dates: First submitted 2023-11-07; First posted 2023-11-22 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Child Wellbeing; Adolescent Health; Quality of Life

STUDY DESIGN:
Intervention Model Description: This study has a quasi-experimental Extended Selection Cohorts (ESC) design. The ESC design is a cohort-longitudinal design with adjacent cohorts, that are measured at two or more time points.
  To separate any effects of the intervention from changes in variables due to other causes, a "wait list control group" element will be applied, i.e., delayed intervention/stepped wedge design: ½ of the schools will start the intervention in November 2023, while the remaining schools will start the intervention in January 2024.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention from November 2023 (Experimental): Pupils in this arm receive the teaching material from November 2023
  Interventions: Behavioral: 5Ways@School
- Wait-list control from November 2023 and intervention from January 2024 (Other): Pupils in this arm constitute a control group from November 2023 until they receive the teaching material from January 2024
  Interventions: Behavioral: 5Ways@School

INTERVENTIONS:
Behavioral: 5Ways@School — The 5Ways@School intervention is a teaching material consisting of five elements; Take notice, Be active, Keep Learning, Connect, and Give. The intervention will be given in an ordinary classroom setting by the class' main teacher in two school hours of 45 minutes each week for six consecutive weeks, i.e., a total of 12 school hours. The teaching sessions will consist of presentations of the five elements, videos, reflection exercises, focused group discussions, creative group work, and giving the pupils small "challenges" to practice what they have learned between the weekly sessions.

SUMMARY:
The aim of this study is to develop a teaching material built on the Five Ways to Wellbeing and investigate its effects on wellbeing and mental health among school pupils aged 10 to 16 years in Moss municipality, Norway. The main questions it aims to answer are:

1. How do participating pupils, teachers, and other school personnel experience the teaching material - is it acceptable and experienced as useful?
2. What are the immediate and long-term effects of the teaching material on the pupils' wellbeing and mental health?
3. For whom is the teaching material effective, and what mechanisms may explain potential improvements in wellbeing after exposure to the teaching material?

Pupils will be given a teaching program at school, delivered by their teacher. Participating pupils and their teachers will be invited to complete questionnaires. Some teachers, school leaders, school health nurses, and parents will be invited to share their experiences with the teaching material in focus group discussions.

DETAILED DESCRIPTION:
Background:

Mental health problems are common among children and adolescents worldwide, and the prevalence of mental distress and common mental disorders has increased in recent years. The recent Coronavirus pandemic has been challenging for the mental health and wellbeing of many children and adolescents; and in Norway higher levels of depressive symptoms and less optimistic future life expectations have been observed among adolescents as a result of the pandemic.The global challenge of mental health problems calls for different approaches; both treating mental health disorders, preventing mental health problems, and promoting mental health and wellbeing for all. School-based interventions are a primary tool in universal prevention to promote mental health and wellbeing, but well-designed interventions with proven long-term effects are rare.

The aim:

The aim of this study is to develop a teaching material built on the Five Ways to Wellbeing and investigate its effects on wellbeing and mental health among school pupils aged 10 to 16 years in Moss municipality, Norway.

The objectives are:

1. To adapt the existing Five ways to wellbeing course for adults to a school setting, and to pilot the intervention in two schools.
2. To explore how participating pupils, teachers, and other school personnel experience the pilot intervention, and identify aspects that should be adjusted before proceeding to a full scale trial.
3. To examine how the teachers deliver the intervention in the full scale trial; their motivation, obstacles they encounter, general satisfaction with the intervention, and their adherence to the intervention manual (i.e., fidelity).
4. To investigate whether the intervention is acceptable and experienced as useful for participating school pupils, parents, teachers, and other school personnel.
5. To investigate whether the intervention have any adverse effects, such as triggering negative emotions.
6. To evaluate the process of implementation.
7. To describe the pupils' wellbeing and mental health at baseline (November 2023).
8. To examine the immediate and long-term effects of the intervention on the pupils' wellbeing and mental health.
9. To assess for whom the intervention is effective (i.e., subgroup analysis and moderation analysis, for example socioeconomic status, gender, and baseline symptom levels).
10. To investigate what mechanisms explain potential improvements in wellbeing after exposure to the interventions.

Sample and recruitment:

Moss municipality has decided to give the "5 Ways@School" teaching material to all pupils aged 10-16 years in the municipality's public schools (n=16) as part of the schools' regular curriculum. In some schools the teaching will start in November 2023 while the remaining schools will start teaching in February 2024, ensuring a "delayed intervention" effect for approximately 50 % of the pupils. All pupils (n=3324) and their teachers (n=156) will be invited to complete questionnaires. The teachers also will be invited to share their experiences with the teaching material in focus group discussions.

Procedures:

The teaching material consists of five elements; Take notice, Be active, Keep Learning, Connect, and Give. The intervention will be given in an ordinary classroom setting by the class' main teacher in two school hours of 45 minutes each week for six consecutive weeks, i.e., a total of 12 school hours. The teaching sessions will consist of presentations of the five elements, videos, reflection exercises, focused group discussions, creative group work, and giving the pupils small "challenges" to practice what they have learned between the weekly sessions. Web-based questionnaires will be administrated and distributed by the PI via the teachers.

Power analysis:

The PI assumes a participation rate of 70 percent among the invited pupils, i.e., approximately 2300 participants. An estimation of statistical power in this study revealed a power of 0.8411 to detect an effect equal to 0.16.

ELIGIBILITY:
Inclusion Criteria:

1. Being a pupil in 5th to 10th grade in a public school in Moss municipality, OR
2. Being a teacher who teaches the Five Ways at School to a school class in one of the participating schools.

Exclusion Criteria: None. However, one school for pupils with special needs (n=18) does not participate in the study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2476 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Change in subjective wellbeing (global life satisfaction - present) | Week 0, 7, 12, 17, and 52
  As a measure of present wellbeing, a version of the Cantril Ladder Scale will be used, one that has been used in the Young in Norway study (Cantril, 1965). Pupils are asked to evaluate their life at the present time, on a scale from 0 (feeling very poor) to 10 (feeling very well).
Change in subjective wellbeing (global life satisfaction - future) | Week 0, 7, 12, 17, and 52
  As a measure of the pupils' expected future wellbeing, a version of the Cantril Ladder Scale will be used, one that has been used in the Young in Norway study (Cantril, 1965). Pupils are asked to estimate how good or bad their life will be in five years from now, on a scale from 0 (feeling very poor) to 10 (feeling very well).
Change in subjective wellbeing (life satisfaction and self-esteem) | Week 0, 7, 12, 17, and 52
  The following measures of life satisfaction and self-esteem will be assessed on a four-point scale ranging from "totally agree" to "totally disagree": "My life is good", "I have all I want in life", "I like myself the way I am", and "I am very satisfied with how I am".
Change in subjective wellbeing (satisfaction with different life domains) | Week 0, 7, 12, 17, and 52
  Satisfaction with the different life domains will be measured by asking the pupils "how satisfied are you with the following aspects of your life: your parents, your friends, your school, your neighborhood, your health, and your appearance?". Pupils respond to each item on a four-point scale ranging from "not at all" to "very satisfied".
Change in social relationships (friends in general) | Week 0, 7, 12, 17, and 52
  Relationships with friends will be assessed by asking the pupils: "Do you have a friend whom you can trust and talk to about everything?", with response options "Yes, I am sure", "Yes, I think so", "I don't think so", and "I have no friends, nowadays".
Change in social relationships (friends during leisure time and school breaks) | Week 0, 7, 12, 17, and 52
  The pupils will be asked two items; "Do you have [a friend] to be with during 1) your leisure time and 2) in the school breaks?" These items will be measured by a four-point scale ranging from "Yes, always" to "No, never".
Change in depressive symptoms | Week 0, 7, 12, 17, and 52
  Depressive symptoms will be measured by Kandel and Davies's six-item Depressive Mood Inventory, assessing depressive symptoms during the preceding week on a four-point scale from 'affected not at all' to 'affected extremely'. In addition, the prosocial items from the Strengths and Difficulties Questionnaire (SDQ) will be used.
Change in loneliness | Week 0, 7, 12, 17, and 52
  Loneliness will be assessed by one item on feelings of loneliness in the past week, on a four-point scale from 'affected not at all' to 'affected extremely'.
Change in leisure activities (time spent per week) | Week 0, 7, 12, 17, and 52
  The respondents' weekly leisure activities will be assessed with the following items: "In your leisure time, how often do you 1) meet with friends in their homes, 2) hang out with friends [outdoor], 3) exercise or do sports, 4) ride a horse, 5) stay at a youth activity club, 6) play an instrument, 7) do things together with your family, 8) help at home doing chores, 9) relax on your own most of the evening". The pupils will respond on a six-point scale ranging from "never" to "every day".
Change in leisure activities and screen time (time spent per day) | Week 0, 7, 12, 17, and 52
  The respondents' daily leisure activities and screen time will be assessed with the following items: "In your leisure time, how many hours a day do you 1) watch tv, tv series, or online videos 2) read books, 3) play computer games, 4) play games on your mobile phone, 5) use social media, 6) read/watch news". The pupils will respond on a six-point scale ranging from "no time" to "3 hours or more".
Acceptability and feasibility 1 (teachers) | Post-intervention at week 7 and 12, respectively
  The teachers will respond on a four-point scale from "agree completely" to "disagree completely" to the following items: "1) I was well motivated to teach the 5Ways@School, 2) I enjoyed teaching the 5Ways@School, 3) Teaching life skills through the 5Ways@School is a natural part of my job as a teacher, 4) I got sufficient information and/or training before I started teaching the 5Ways@School, 5) I think the pupils learned something new and useful, 6) There was too little activities in the 5Ways@School, 7) There was too much activities in the 5Ways@School, 8) I followed the teaching manual to a high degree, 9) I completed all the six lessons in the 5Ways@School, 10) I had to abbreviate one or more lesson(s), 11) I think that the 5Ways@School should be part of the ordinary school curriculum in 5h to 7th grade, and 12) I think that the 5Ways@School should be part of the ordinary school curriculum in 8th to 10th grade."
Acceptability and feasibility 2 (teachers) | Post-intervention at week 7 and 12, respectively
  The teachers who will be teaching the interventions will be asked: "Based on your experiences, which of the five elements in the 5Ways@School do you think was 1) most useful for the pupils?, easiest for you to teach, and 3) most challenging for you to teach?" The teachers will respond to these questions by choosing any of the five elements of the 5Ways@School: Take notice, Be active, Keep Learning, Connect, and Give.
Acceptability and feasibility 3 (pupils) | Post-intervention at week 7 and 12, respectively
  The pupils will be given a questionnaire with the following items: "1) I enjoyed learning about 5Ways@School, 2) I learned something new, that I can make use of, 3) The teaching was easy to understand, 4) The teaching was boring, 5) The teaching was interesting, 6) There was too little activities, 7) There was too much activities, 8) The teaching made me sad, afraid, or angry, 9) The teaching made me happy, 10) I will practise more of the five ways in the future, 11) I think all pupils should learn about the five ways." The pupils will respond on a four-point scale from "agree completely" to "disagree completely"

SECONDARY OUTCOMES:
Socio-economic status | Week 0 and 17
  Family socio-economic status will be assessed by a composite score four items from the Health Behaviour in School-Aged Children (HBSC) Family Affluence Scale (Currie et al., 1997, 2008), which include frequency of traveling for family holidays in the previous year, number of computers and cars in the family, and the participant having an individual room at home. The scale ranges from 0 to 9, where a low score indicates low socio-economic status.
Other demographics | Week 0 and 17
  Gender will be assessed. Only school grade (grades 5 to 10) but not age will be assessed. The pupils will be asked whether both their parents are born in a country other than Norway, and whether they have one or two homes.
Pupils' knowledge of other health promoting programs | Post-intervention at week 7 and 12, respectively
  Pupils will be asked whether their class/school has completed one of the following teaching programs: 1) "Sam", and 2) "Robust Youths". Response options are "yes" and "no".

CONTACTS AND LOCATIONS:
Overall Officials: Ragnhild B Nes, PhD, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Kristian Green Krogshus, Moss, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krogshus KG, Bjertness E, Czajkowski NO, Rodriguez-Cano R, Nes RB. Study protocol for 5Ways@School - An implementation and effectiveness trial of a school-based wellbeing intervention in 16 schools in Norway. Scand J Public Health. 2025 Sep 8:14034948251370109. doi: 10.1177/14034948251370109. Online ahead of print. PMID 40916894
- See also: Information on Moss municipality's homepage (in Norwegian) — https://www.moss.kommune.no/alle-tjenester/horinger-planer-og-prosjekter/kommunens-prosjekter-utviklingsarbeid-og-forskning/kommunens-utviklingsarbeid-og-forskning/prosjekt-fem-gode-vaner-hverdagsglede-skole/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT06144502/Prot_SAP_002.pdf